CLINICAL TRIAL: NCT01761877
Title: NSAID Effects on Clinical and Imaging Breast Biomarkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Alison Stopeck, Professor, Stony Brook University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1RO1 CA1615301A1; 12-0080-04 (Other: UArizona); 676847 (Other: Stony Brook University)
Record Dates: First submitted 2012-12-28; First posted 2013-01-07 (Estimated); Results first posted 2023-02-10 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-01

CONDITIONS: Inflammation; Cancer; Pain; Hypertension
Keywords: breast cancer, breast density, chemoprevention
MeSH Terms: conditions — Inflammation; Neoplasms; Pain; Hypertension; Breast Neoplasms | interventions — Sulindac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sulindac (Clinoril) (Experimental): Women taking aromatase inhibitors for adjuvant therapy for their breast cancer will receive 150 mg of sulindac twice daily for 12 months. They will receive up to 4 MRI within 12 months.
  Interventions: Drug: Sulindac
- Observational (No Intervention): Women taking aromatase inhibitors for adjuvant therapy for their breast cancer will continue their treatment will be monitored with MRI and standard of care tests every 6 months for up to 12 months.

INTERVENTIONS:
Drug: Sulindac
  Other Names: Clinoril
  Arms: Sulindac (Clinoril)

SUMMARY:
This study has two purposes. One is to determine if daily sulindac decreases breast density; a risk factor for breast cancer development. The second is to determine whether sulindac reduces pain and stiffness associated with regular use of aromatase inhibitors given for the treatment of breast cancer.

DETAILED DESCRIPTION:
To accomplish our study aims, we will conduct a phase II, single are trial of sulindac in postmenopausal women with early stage ER+ breast cancer who are receiving an aromatase inhibitor as adjuvant hormonal therapy. Approximately 75 breast cancer patients, stable on AI therapy (minimum of 3 months) for the treatment of their breast cancer will receive sulindac 150 mg bid for 12 months. Breast imaging will be conducted at baseline, 6 and 12 months.

The primary endpoint of the study will be change in the appearance of the contralateral, uninvolved breast as measured by quantitative Fat Water Ratio (FWR-MRI) mapping at 12 months in response to sulindac therapy. As changes in breast density in the contralateral, uninvolved breast will be the primary endpoint of the study, patients with bilateral breast cancer or those patients undergoing bilateral mastectomies or reconstruction surgery will be ineligible. Secondary endpoints of the trial include 12 month change in general pain and joint specific stiffness and pain as assessed by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). A number of exploratory endpoints are planned and include comparison of MRI measures of the breast, tissue biomarkers, and pain at 6 months as early indicators of 12 month responses. For the tissue biomarkers, core needle biopsies will be obtained in a subset of women who consent to the procedure from the uninvolved contralateral breast at baseline and at 6 months. Tissue studies will include characterization of tissue histology (graded by cellularity and stromal elements) and molecular measures of proliferation and apoptosis.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria will include: Postmenopausal women with of first incidence of early stage (stages 0 - III) hormone receptor positive breast cancer stabilized on anastrozole therapy for at least 3 months
* Patients must have started on anastrozole and plan to continue on anastrozole therapy for a minimum of 12 months
* Patients must have an unaffected, non-irradiated contralateral breast with a baseline breast density score of > 25% as measured by standard digital mammography (BIRADs score > 2) or magnetic resonance imaging (MRI) performed within 12 months of randomization to the study
* A willingness to follow the study protocol, as indicated by provision of informed consent to participate
* A willingness to avoid taking NSAIDs outside of the trial (rare NSAID use for musculoskeletal symptoms excepted)
* Normal renal function as determined by a serum creatinine < upper limit of normal
* No known contraindication to NSAID use
* Normotensive or controlled blood pressure (< 140/90) on a single anti-hypertensive medication

Exclusion Criteria:

* Current or anticipated need for daily aspirin or NSAID use including aspirin for cardiovascular protection
* Known intolerance to NSAIDs
* Age > 75 years
* History of cardiovascular disease including prior myocardial infarction, angina, stroke, or transient ischemic attack (TIA)
* Diabetes requiring drug therapy
* Current smoker
* History of Uncontrolled hypertension
* Blood pressure > 140/90 at baseline by home monitoring
* History of GI ulcers, chronic GERD, or GI bleeding in the past 5 years
* History of a bleeding diathesis or current anticoagulant therapy
* Daily therapy with H2 blockers or protein pump inhibitors
* History of claustrophobia
* Have electrically, magnetically, or mechanically activated implants including cardiac pacemaker, cochlear implants, magnetic surgical clips or prostheses.

Max Age: 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-12; Primary Completion 2019-02-07 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Thompson-Carino, PhD, Principal Investigator — Stony Brook University; Alison Stopeck, MD, Principal Investigator — Stony Brook University; Pavani Chalasani, MD, Principal Investigator — University of Arizona
Locations (2):
- United States (2):
  - University of Arizona Cancer Center, Tucson, Arizona
  - Stony Brook University Cancer Center, Stony Brook, New York

REFERENCES:
- [Derived] Martinez JA, Wertheim BC, Roe DJ, Chalasani P, Cohen J, Baer L, Chow HS, Stopeck AT, Thompson PA. Sulindac Improves Stiffness and Quality of Life in Women Taking Aromatase Inhibitors for Breast Cancer. Breast Cancer Res Treat. 2022 Feb;192(1):113-122. doi: 10.1007/s10549-021-06485-0. Epub 2022 Jan 18. PMID 35039952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients were enrolled at the University of Arizona Cancer Center and at the Stony Brook Cancer Center.
Pre-assignment Details: Patients assigned to receive sulindac were required to complete a NSAID washout period.
Groups:
- Sulindac (Clinoril): Women taking aromatase inhibitors for adjuvant therapy for their breast cancer will receive 150 mg of sulindac twice daily for 12 months. They will receive up to 4 MRI within 12 months.
  Sulindac
- Observational: Women taking aromatase inhibitors for adjuvant therapy for their breast cancer will continue their standard of care treatment and be monitored with MRI for change in breast density every 6 and 12 months.
Period: Overall Study
Arm/Group | Sulindac (Clinoril) | Observational
Started (A total of 58 patients enrolled and initiated a 4-month NSAID washout, of which 50 started sulindac treatment and 43 completed to 12 months.) | 58 | 56 (A total of 56 patients enrolled to observation but 6 withdrew or became ineligible before their baseline MRI.)
Completed | 43 | 40
Not Completed | 15 | 16
Not completed — Adverse Event | 7 | 0
Not completed — Withdrawal by Subject | 6 | 4
Not completed — Stopped taking AI Aromatase Inhibitor | 1 | 5
Not completed — Death | 0 | 1
Not completed — MRI intolerant | 1 | 6

BASELINE CHARACTERISTICS:
Population: For baseline analyses for the sulindac arm, we included only those participants who remained in the study after the NSAID washout and who started the intervention with sulindac (n=50). For the baseline analyses for the observation arm, we included those participants who either completed their baseline MRI and/or questionnaires for the secondary arthralgia endpoints (n=50).
Groups:
- Observational: Women taking aromatase inhibitors for adjuvant therapy for their breast cancer will continue their treatment and will be monitored with MRI and standard of care tests at 6 and 12 months.
- Total: Total of all reporting groups
Arm/Group | Sulindac (Clinoril) | Observational | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (5.5) | 64.2 (6.6) | 63.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, Non-Hispanic | 44 | 46 | 90
  Black, Non-Hispanic | 1 | 0 | 1
  Hispanic | 3 | 3 | 6
  Asian, Non-Hispanic | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in Breast Density Measured as Fat to Water Ratio by Magnetic Resonance Imaging
Description: Adjusted estimates of relative change in percent breast density by magnetic resonance imaging
Time Frame: Baseline and 12 months
Population: Breast density data were unavailable for 4 participants in the observation group due to MRI intolerance. This reduced the sample size for the outcome of change in breast density for the observation arm compared to the secondary endpoints.
Measure: Mean (95% Confidence Interval); unit: percent change in breast density
Groups:
- Observational: Women taking aromatase inhibitors for adjuvant therapy for their breast cancer will continue their treatment and will be monitored with MRI and standard of care every 6 months for up to 12 months.
Arm/Group | Sulindac (Clinoril) | Observational
Number analyzed (Participants) | 50 | 46
percent change in breast density | -9.8 [-14.6 to -4.7] | -3.6 [-8.9 to 2.0]
Statistical Analysis 1: Comparison: Sulindac (Clinoril) vs Observational; The study was designed to assess change in breast density using fat/water MRI after 12 months of sulindac intervention in postmenopausal breast cancer patients taking aromatase inhibitors for the treatment of estrogen receptor positive breast cancer. A non-randomized observation arm was included with the same eligibility criteria to assess change in breast density over 12 months using the fat/water MRI method of quantifying breast density. Change was examined separately for each arm; Test type: Other — Mixed Models Analysis; p < 0.05, Mixed Models Analysis — A p value was calculated for change in breast density from baseline to 12 months separately for each study arm

2. Secondary Outcome: Muscle and Joint Pain and Stiffness
Description: The endpoint for arthralgia is change from baseline in Total Western Ontario and McMaster Universities Osteoarthritis (WOMAC) Index scores on a scale at 12 months. The Western Ontario and McMaster Universities Index is a self-administered questionnaire consisting of 24 items divided in 3 subscales: Pain, Stiffness, and Physical Function. Scores on the scale range from 0 to 96 for total WOMAC where 0 represents the best health status and 96 the worst possible status.
Time Frame: Baseline and 12 months
Population: Questionnaires for patient reported outcomes were completed at baseline for 50 participants in both sulindac and the observation group.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Sulindac (Clinoril) | Observational
Number analyzed (Participants) | 50 | 50
score on a scale | -5.85 [-9.73 to -1.96] | -0.25 [-3.25 to 2.69]
Statistical Analysis 1: Comparison: Sulindac (Clinoril) vs Observational; Test type: Other; p < 0.05, Mixed Models Analysis — A p value of <0.05 was selected for change in each arm. The study did not include a direct comparison between the two arms

3. Other Pre Specified Outcome: Change in Mean Arterial Blood Pressure at 12 Months
Description: Adjusted estimate of change in mean arterial blood pressure in each study arm at 12 months in each study arm.
Time Frame: Change in blood pressure between Baseline and 12 months
Population: Blood pressure was available at baseline for 50 participants in both the sulindac and observation group.
Measure: Mean (95% Confidence Interval); unit: mm Hg
Groups:
- Sulindac: Women taking aromatase inhibitors for adjuvant therapy for their breast cancer will receive 150 mg of sulindac twice daily for 12 months.
Arm/Group | Sulindac | Observational
Number analyzed (Participants) | 50 | 50
mm Hg | 0.77 [-1.82 to 3] | 1.52 [-1.17 to 4]
Statistical Analysis 1: Comparison: Sulindac vs Observational; Test type: Other; p < 0.05, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 13 months.
Description: Participants in the observation only group were not systematically followed for adverse events. There was not active intervention and there was not intent to compare the two groups.
Groups:
- Sulindac (Clinoril): Women taking aromatase inhibitors for adjuvant therapy for their breast cancer will receive 150 mg of sulindac twice daily for 12 months. They will receive up to 4 MRI within 12 months and two breast biopsies.
Arm/Group | Sulindac (Clinoril) | Observational
All-Cause Mortality (participants affected / at risk) | 0/50 | 1/50
Serious Adverse Events (participants affected / at risk) | 3/50 | 1/50
Other Adverse Events (participants affected / at risk) | 25/50 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulindac (Clinoril) (N=50) | Observational (N=50)
Intraparenchymal Hemorrhage associated with cerebral amyloid angiopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient Pancreatitis of Unclear Etiology (Gastrointestinal disorders) | 1 (1) | 0 (0)
B cell Lymphoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Antral Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sulindac (Clinoril) (N=50) | Observational (N=0)
upset stomach or pain (Gastrointestinal disorders) | 6 (6) | 0 (0)
rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
headache (Nervous system disorders) | 3 (3) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
hypertension (Vascular disorders) | 7 (7) | 0 (0)
insomnia (Psychiatric disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT01761877/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-04): https://cdn.clinicaltrials.gov/large-docs/77/NCT01761877/SAP_001.pdf